CLINICAL TRIAL: NCT03191201
Title: A Double Blind Randomised Placebo-controlled Trial to Assess the Effect of a Single Administration of Ferric Carboxymaltose of 1000 mg Iron on Glucose Homeostasis, in Iron-deficient Non-anaemic Women of Childbearing Age.
Brief Title: A Double Blind Randomised Placebo-controlled Trial to Assess the Role of Iron Repletion in Glucose Homeostasis.
Acronym: DIAFER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The reason for early termination is difficulties recruiting that caused a premature ending of financial resources ensuring protected time for research.
Sponsor: Prof Gérard WAEBER (Other)
Collaborators: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); Centre Hospitalier Universitaire Vaudois (Other); University of Lausanne (Other)
Responsible Party: Sponsor-Investigator, Prof Gérard WAEBER, Head of the Department of Medicine, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016-01449
Record Dates: First submitted 2017-05-17; First posted 2017-06-19 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Iron-deficiency; Iron Toxicity; Glucose Metabolism Disorders (Including Diabetes Mellitus); Metabolic Side Effects of Drugs; Metabolic Disorder, Glucose; Safety Issues
Keywords: Metabolomics, Transcriptomics, Ironomics
MeSH Terms: conditions — Anemia, Iron-Deficiency; Glucose Metabolism Disorders; Metabolic Side Effects of Drugs and Substances | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double blind randomised placebo-controlled, parallel group comparative inferiority study with open-label extension divided in two parts:
  * A first randomised and double-blind part in which FCM or placebo will be administered at baseline and post-baseline parameters assessed.
  * A second non-randomised, non-blinded open-label extension part starting at the end of part 1, in which participants randomised to the placebo group will receive a FCM injection and post-baseline parameters assessed.
Who Masked: Participant, Outcomes Assessor
Masking Description: To ensure that patients are unaware of the study drug they are receiving, the infusion pouch will be prepared in a separate room by members of the pharmacy unit and opaque bags will cover the infusion kits and infusions will be done via dark coloured infusion sets. Finally, a curtain will be used to shield the injection site from the patient's view.
  To ensure that Outcomes Assessors are unaware of the study drug the patient is receiving, a seperate team of care providers will supervise the infusion of the investigation product and collect and/or manage adverse events (AEs) and serious adverse events (SAEs). The Outcome Assessor will not have access to participant related data during the randomised part of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric carboxymaltose arm (Active Comparator): Ferric carboxymaltose (FCM), 1000 mg iron element will be administered once by drip infusion (Intravenous route). FCM will be diluted in 250 mL of a commercially available sterile 0.9% sodium chloride solution prior to administration. Infusion time will be 15 minutes.
  Interventions: Drug: Ferric Carboxymaltose
- Placebo arm (Placebo Comparator): A commercially available sterile, 250 mL, 0.9% sodium chloride solution will be administered by drip infusion (Intravenous route). Infusion time will be 15 minutes.
  At the end of the randomised part of the study, participants initially randomised to the placebo group will be included in a non-blinded open-label extension part and receive a FCM 1000 mg injection.
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: Ferric Carboxymaltose — Ferric Carboxymaltose 1000 mg iron element will be diluted in 250 mL of a commercially available sterile 0.9% sodium chloride solution.
  Arms: Ferric carboxymaltose arm
Drug: 0.9% sodium chloride solution — 250 mL of a commercially available sterile 0.9% sodium chloride solution.
  Arms: Placebo arm

SUMMARY:
In this study the investigators aim at addressing potential relationships between iron stores and glucose homeostasis. Iron (i.e. Ferric Carboxymaltose) will be perfused to pre-menopausal, iron-deficient non-anaemic women suffering from a chronic fatigue syndrome and parameters related to glucose homeostasis, parameters related to metabolic syndrome and inflammation will be measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women.
* Negative pregnancy test.
* Adequate contraception during the study period and for 1 month following study completion.
* Overt or relative iron deficiency at screening defined as follows:

Serum ferritin <50 ng/mL AND transferrin saturation <20%, OR Serum ferritin <30 ng/mL.

- Serum C-reactive protein: <5 mg/L if not on oral contraception, OR <20 mg/L if use of oral contraception

* Intolerance to oral iron formulations, or lack of efficacy of oral iron formulations.
* Minimum total score of 5 on the Visual analogic scale of fatigue.
* Normal levels of vitamin B12 and folic acid at screening.
* Availability and willingness to complete all study visits and procedures per protocol.
* Ability to sign an informed consent.

Exclusion Criteria:

* Age <18 years.
* Menopause (defined as an amenorrhea of at least 12 months).
* Irregularly menstruating women (menstrual cycle outside a range of 24-38 days in duration) or experiencing overt metrorrhagia (simple spotting not being an exclusion criteria).
* Body mass index <18.5 kg/m2 or >30 kg/m2.
* Diabetes, defined as subjects with HbA1c ≥ 6.5 % and/or with fasting blood glucose levels ≥ 7 mmol/l and/or with a history of diabetes and/or by the use of anti-diabetic drugs.
* Hb level <117 g/L or known haemoglobinopathy or haemochromatosis.
* Blood transfusion within the last 12 weeks.
* Intake of iron preparations 4 weeks prior to screening.
* Known hypersensitivity to FCM or to any other iron preparation.
* Suspicion of major depressive disorder based on Patient Health Questionnaire.
* Known chronic inflammatory disease, including human immunodeficiency virus, hepatitis B or hepatitis C virus infection.
* Active malignancy.
* Decreased renal function (estimated glomerular filtration rate using the CKD-EPI equation<60 ml/min/1.73m2).
* Liver dysfunction (aspartate aminotransferase and alanine aminotransferase > 3-fold upper limit).
* Angina (Class IV).
* Asthma.
* Documented sleep apnoea.
* Important recent weight loss (>10% within the past month).
* Thyroid dysfunction (thyroid stimulating hormone >4 µU/mL).
* Reported weekly alcohol consumption > 14 standard drinks.
* Drug abuse (any drug consumption reported in the past 12 months).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glucose homeostasis status, assessed by a dynamic two-step hyperglycaemic clamp investigation. | at 28 days of the injection of the Investigation Product
  two-step hyperglycaemic clamp investigation

SECONDARY OUTCOMES:
Change from baseline in ultrasensitive C-reactive protein (hs-CRP) levels at 14 days | at 14 days of the injection of the Investigation Product
  plasma hs-CRP levels
Change from baseline in ultrasensitive C-reactive protein (hs-CRP) levels at 28 days | at 28 days of the injection of the Investigation Product
  plasma hs-CRP levels
Change from baseline in interleukin-6 (IL-6) levels at 14 days | at 14 days of the injection of the Investigation Product
  plasam IL-6 levels
Change from baseline in interleukin-6 (IL-6) levels at 28 days | at 28 days of the injection of the Investigation Product
  plasam IL-6 levels
Change from baseline in adiponectin levels at 14 days | at 14 days of the injection of the Investigation Product
  adiponectin
Change from baseline in adiponectin levels at 28 days | at 28 days of the injection of the Investigation Product
  adiponectin
Change from baseline in interleukin-1beta levels at 14 days | at 14 days of the injection of the Investigation Product
  IL-1b
Change from baseline in interleukin-1beta levels at 28 days | at 28 days of the injection of the Investigation Product
  IL-1b
Change from baseline in blood pressure levels at 14 days | at 14 days of the injection of the Investigation Product
  systolic and diastolic blood pressure
Change from baseline in blood pressure levels at 28 days | at 28 days of the injection of the Investigation Product
  systolic and diastolic blood pressure
Change from baseline in the plasma lipid profile level at 14 days | at 14 days of the injection of the Investigation Product
  plasma total- and HDL-cholesterol and plasam triglycerides
Change from baseline in the plasma lipid profile level at 28 days | at 28 days of the injection of the Investigation Product
  plasma total- and HDL-cholesterol and plasam triglycerides
Change from baseline in the Homeostasis Model Assessment (HOMA-2) index at 14 days | at 14 days of the injection of the Investigation Product
  Calculated Homeostasis Model Assessment (HOMA-2) index
Change from baseline in the Homeostasis Model Assessment (HOMA-2) index at 28 days | at 28 days of the injection of the Investigation Product
  Calculated Homeostasis Model Assessment (HOMA-2) index

OTHER OUTCOMES:
Change from baseline in the plasma metabolomic profiling as assessed by metabolomics | at 14 and 28 days of the injection of the Investigation Product
  Metabolomics
Change from baseline in circulating miRNAs | at 14 and 28 days of the injection of the Investigation Product
  selected miRNA as measured by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Waeber, MD, Study Director — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (1):
- Policlinique Médicale Universitaire, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaccard E, Seyssel K, Gouveia A, Vergely C, Baratali L, Gubelmann C, Froissart M, Favrat B, Marques-Vidal P, Tappy L, Waeber G. Effect of acute iron infusion on insulin secretion: A randomized, double-blind, placebo-controlled trial. EClinicalMedicine. 2022 May 6;48:101434. doi: 10.1016/j.eclinm.2022.101434. eCollection 2022 Jun. PMID 35706490